CLINICAL TRIAL: NCT05500833
Title: Multidimensional Characterization of Dyspnea in Children
Acronym: DYSPED
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220874
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Dyspnea and Respiratory Insufficiency in Children
Keywords: Dyspnea; Multidimensional; chidren; chronic respiratory insufficiency; acute respiratory insuffisciency; multidimensional dyspnea profile; respiratory distress observation scale
MeSH Terms: conditions — Dyspnea | interventions — dipeptidase 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Multidimentional observation scale (MDP) — Upon arriving to the hospital (for an hospitalization or a consultation), a trained and declared investigator will inform the patients and their parents of the study, orally and using a written information note. Participation to the study will also be proposed to under aged children in an adequate language and a specific information note will be handed to them. If they wish, they will have a 20 min reflexion time before deciding on participating to the study.One the patient is included, the study will unfold as follows. First, Evaluation of acute dyspnea: general data and dyspnea scores will be collected upon inclusion, and dyspnea score will be collected once again 30 min later, and subsequently one a day until the end of hospitalization (test-retest). Data from clinical examination and treatment modifications will also be collected daily. Second, Evaluation of chronic dyspnea: general data and dyspnea scores will be collected upon inclusion and 1 to 1.5h later
  Other Names: Respiratory distress observation scale (RDOS)

SUMMARY:
There is no specific tool existing to describe dyspnea in children in a multidimensional way.

It has been shown in adult studies that multidimensional dyspnea evaluation scales are well correlated to quality of life and respiratory function impairments.

The investigators hypothesis is that using multidimensional dyspnea evaluation scales could allow for a more systematic and precise evaluation of this symptom in children, thus improving management and follow-up of patients presenting with acute (asthma attack, infectious diseases) and chronic (cystic fibrosis, primary ciliary diskynesia, neuromuscular diseases) respiratory insufficiency.

DETAILED DESCRIPTION:
Introduction Breathing is most of the time an activity realized ion an automated way. In various situations however, it can be "felt", for example when people are producing an effort. To term used to refer to these situation is "breathlessness". When breathing is perceived as an unpleasant sensation, causing suffering, especially in the context of diseases that are often of cardiac or respiratory origin, the appropriate term is "dyspnea".

In 1999, a consensus conference defined dyspnea as a subjective experience of respiratory discomfort consisting in sensations of distinct quality and varying intensity.

Sensory and emotional aspects associated to dyspnea have been compared to those observed in pain. Pain is often defined according to its intensity, quality and temporal evolution of its sensory dimension, but also according to the emotional response it induces. There are similarities between pain and dyspnea, two unpleasant sensations sharing common physiological substrates. Two studies have previously demonstrated that there is an overlap between cerebral regions activated during pain and those activated when dyspnea occurs. This is in favor of analyzing dyspnea according to the same sensory and emotional dimensions as pain.

To those intrinsic sensory characteristics are added psychological, social and economic factors that may have an influence, positively or negatively, on the sensation of dyspnea.

Scientific background Dyspnea is multifactorial and multidimensional. Its multidimensional nature can be apprehended using specific tools and questionnaires designed to this effect. Among them, the Dyspnoea-12, the Multidimensional Dyspnea Profile (MDP) ans the Respiratory Distress Observation Scale (RDOS). These scales take into account not only the intensity of dyspnea, but also its sensory qualities and affective dimension, which can vary independently from one another. All these scales have already been validated in French language.

The RDOS The RDOS is an hetero-questionnaire divided in 8 items: respiratory rate, heart rate, restlessness (non-purposeful movements), accessory muscle use (rise in clavicule during inspiration), grunting at end-expiration (guttural sound), Nasal flaring (involuntary movement of nares) and look of fear. Each item is scored between 0 (absence) and 2 (presence) points.

The MDP The MDP, which has already been validated in French speaking language, is a self report questionnaire including 11 items, each one evaluated by a scale ranging from 0 to 10, describing the intensity, sensory and emotional characteristics of dyspnea. The MDP score can be analyzed in terms of immediate perceptual response, emotional response or affective dimension, similarly to models applied to pain.

The MDP isn't defendant on physiological variables changing with age that is why the scale validated in adults will be used for children aged between 12-18 years. A simplified MDP will be used for children aged between 6-12 years.

RDOS and MDP in the clinical set-up In adults, the MDP has previously been used to evaluate dyspnea in patients with chronic bronchopulmonary dysplasia (COPD) or Amyotrophic lateral sclerosis (ALS). Is has allowed a better comprehension of the impact of dyspnea on patients' quality of life. It has also been used to evaluate the efficacy of various therapeutic interventions, such as respiratory rehabilitation in COPD patients.

However, the MDP requests adequate communication skills and mastering the vocabulary. This is an obstacle in younger children and, more broadly, in non-communicative patients. The RDOS has been develop to allow an hetero-evaluation of dyspnea in palliative care patients unable to communicate and describe their symptoms. This scale has also demonstrated A good correlation to the visual analogue scale-dyspnea and with the clinical evolution of patients in palliative care.

This scale has latter been adapted to patients un intensive care (IC-RDOS) and mechanically ventilated patients (MV-RDOS). It could easily be used in children; however, physiological variables used in the RDOS would need to be adapted to different age groups. A RDOS-infant score has recently been developed for newborns, including the observation of inter-costal and supra-sternal retractions, cyanosis and capillary perfusion. Once more, this score has been developed for newborns only. Moreover, it does not take into account the observation of fearful expressions which could be an important parameter in the evaluation of dyspnea in older children.

Dyspnea in children Various diseases can be responsible for chronic respiratory insufficiency and cause chronic dyspnea, among them cystic fibrosis, primary ciliary dyskinesia, interstitial lung diseases and neuromuscular diseases.

Acute dyspnea is also a frequent cause of hospitalizations, especially when secondary to acute respiratory infections, asthma attacks or acute decompensation of a chronic respiratory disease. Dyspnea can be evaluation by the VAS-dyspnea. In asthmatic patients, it has been shown that this scale allows a good evaluation of bronchial constriction and a good sensitivity to therapeutic interventions. The childhood asthma score (CAS) and preschool respiratory assessment measure (PRAM) score are also commonly used to evaluate the severity of asthma attacks. However, they are unidimensional scales only validated for asthmatic children.

There is no existing scale validated in children providing a multidimensional evaluation of dyspnea, whether it be acute or chronic.

Dyspnea-VAS can be used, but it is a unidimensional scale which does not allow the evaluation of dyspnea's sensory and affective dimensions.

Hypothesis is that using multidimensional evaluation scales for dyspnea, such as the MDP, simplified MDP and RDOS could allow for a reliable evaluation of dyspnea in children aged between 6-18 years.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 6-17 years old at inclusion
* Experiencing respiratory complaints at inclusion
* Social security number
* Children whom parents or legal representatives are present or reachable via phone call at inclusion
* Non-opposition of parents or legal representatives to participate in the study
* Children who are followed at or hospitalized in Trousseau hospital's pediatric pulmonology department for: asthma attack, acute respiratory insufficiency, acute exacerbation of a chronic respiratory disease, chronic respiratory insufficiency.
* For the study of acute dyspnea: patients hospitalized for acute respiratory disease since less than 72h.
* For the study of chronic dyspnea: children presenting with chronic respiratory disease.

Exclusion Criteria:

* Cognitive disorders making it impossible to understand self-assessment scales
* Refusal of the child to participate in the research

For the assessment of chronic dyspnea:

* Children followed for a chronic respiratory pathology having presented an episode of acute respiratory decompensation in the 6 weeks preceding inclusion.

Ages: 6 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Children aged 6 to 17 years old and presenting an acute or chronic respiratory pathology.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2028-02-26 (Estimated); Study Completion 2028-02-26 (Estimated)

PRIMARY OUTCOMES:
Validate the Multidimensional Dyspnea Profale (MDP) self-evaluation scale in children aged between 12 and 17 years presenting with acute or chronic dyspnea. | through study completion, an average of 36 months
  Use of the MDP questionnaire and test if usable and compliant for the teenager. (Scale from 0 to 10, with 10 corresponding to significant breathing difficulties.)

SECONDARY OUTCOMES:
Validate the Respiratory Distress Observation Scale (RDOS) hetero-evaluation scale in patients aged between 12-17 years presenting with acute dyspnea. | through study completion, an average of 36 months
  Use of the RDOS questionnaire to describe dyspnea of teenager (Scale from 0 to 16: 0 = no dyspnea, 16 = maximum dyspnea)
Provide a multidimensional description of dyspnea using the MDP scale in children aged 12-17 y/o. | through study completion, an average of 36 months
  Describe dyspnea of teenager thanks to MDP scale. (Scale from 0 to 10, with 10 corresponding to significant breathing difficulties)
Study the correlation between MDP and RDOS scores and Dyspnea-visual analogue scale (VAS). | through study completion, an average of 36 months
  Compare Multidimensional Dyspnea Profale (MDP, Scale from 0 to 10, with 10 corresponding to significant breathing difficulties.) self-evaluation scale, Respiratory Distress Observation Scale (RDOS, Scale from 0 to 16: 0 = no dyspnea, 16 = maximum dyspnea) scores and Dyspnea-visual analogue scale (VAS, Scale of 0 to 10, a score of 10 corresponds to severe pain)
Validate the use of a simplified MDP in children aged between 6-11 y/o presenting with acute or chronic dyspnea. | through study completion, an average of 36 months
  Use of the Multidimensional Dyspnea Profale (MDP) questionnaire (Scale from 0 to 10, with 10 corresponding to significant breathing difficulties) and test if usable and compliant for the children
Provide a multidimensional description of dyspnea in children aged between 6-11 y/o. | through study completion, an average of 36 months
  Describe results from EVA dyspnea a vertical visual analogue scale as a measure of clinical dyspnea. (Scale from 0 to 10, with 10 corresponding to significant breathing difficulties.)
Study the correlation between the simplified MDP and the dyspnea-VAS. | through study completion, an average of 36 months
  Compare Multidimensional Dyspnea Profale (MDP) questionnaire (Scale from 0 to 10, with 10 corresponding to significant breathing difficulties) and Dyspnea-visual analogue scale (VAS, Scale of 0 to 10, a score of 10 corresponds to severe pain).
Study the association between dyspnea scores and different clinical features, the use of treatments and results of explorations | through study completion, an average of 36 months
  Describe association between different factors
Study the impact of dyspnea on quality of life using the PedSQL scale in children presenting with chronic dyspnea and their families. | through study completion, an average of 36 months
  Describe the impact of dyspnea on quality of life thanks to Paediatric Quality of Life (PedSQL, Scale of 0 to 100, a score of 100 corresponds to a very degraded quality of life due to the disease).
Study the correlation between dyspnea scores in children and their parents' anxity scores using the State-Trait Anxiety Inventory (STAI-Y) questionnaire. | through study completion, an average of 36 months
  Compare between dyspnea scores in children and their parents' anxity scores using the STAI-Y questionnaire (Scale of 0 to 100, a score of 100 corresponds to high anxiety)

CONTACTS AND LOCATIONS:
Locations (1):
- Service de pneumologie pédiatrique, Hôpital Armand Trousseau, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided